CLINICAL TRIAL: NCT01624051
Title: A Phase II Double Blind Randomized Trial Comparing Standard Dosing Based on Body Surface Area Versus Dosing Based on Personalized Lean Body Mass in Patients With Stage IIIB or IV Non-Small Cell Lung Cancer Receiving First Line Cisplatin Based Chemotherapy
Brief Title: A Study Comparing Chemotherapy Dosing Based on Either Standard Body Surface Area or Lean Body Mass in Patients With Advanced Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sawyer - Lung - CCI
Record Dates: First submitted 2012-04-26; First posted 2012-06-20 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Lung Cancer
Keywords: cisplatin based chemotherapy; non-small cell lung cancer; lean body mass; sarcopenia
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Sarcopenia | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Body Surface Area Dosing (Active Comparator): Standard dosing arm based on body surface area
  Interventions: Other: Standard dosing method arm: Cisplatin (chemotherapy) dosing based on body surface area
- Lean Body Mass Dosing (Experimental): Experimental dosing arm based on individual lean body mass
  Interventions: Other: Experimental dosing method arm: Cisplatin (chemotherapy) dosing based on individual lean body mass

INTERVENTIONS:
Other: Standard dosing method arm: Cisplatin (chemotherapy) dosing based on body surface area — Cisplatin dosing calculated at the rate of 75 mg/m2
  Arms: Body Surface Area Dosing
Other: Experimental dosing method arm: Cisplatin (chemotherapy) dosing based on individual lean body mass — Cisplatin dosing calculated at the rate of 3.10 mg/kg lean body mass
  Arms: Lean Body Mass Dosing

SUMMARY:
Cancer patients are highly variable in their body composition, specifically in the proportion of fat and muscle. Some patients tend to gain fat and lose muscle (or lean body mass) at the same time. These patients can develop severe muscle wasting, termed sarcopenia. Patients with sarcopenia have more severe treatment related toxicity requiring delays, dose reductions and stopping of treatment, and have reduced survival. One potential explanation for this is that patients with sarcopenia have a reduced volume of lean body mass into which chemotherapy drugs are distributed, resulting in a higher concentration and greater toxicity. This study will randomize lung cancer patients to either the standard dosing strategy based on body surface area or experimental, personalized dosing based on lean body mass. Based on retrospective findings in this patient population, the investigators expect to find that severe toxicity will be reduced for sarcopenic patients on the personalized dosing arm based on lean body mass.

DETAILED DESCRIPTION:
Retrospective findings of NSCLC patients treated with a cisplatin based chemotherapy regimen show that although all were given cisplatin at the standard rate of 75 mg/m2 according to lean body mass, when this was expressed in relation to individual lean body mass, there was a high degree of variation. Incidence of dose limiting toxicity was 41% in patients whose dose was within + 25% of the median value. However, sarcopenic patients received on average a 35% higher dose and 80% of these patients experienced severe toxicity requiring dose reduction or termination of therapy, a clinically unacceptable level. The relatively muscular subset of patients with higher lean body mass had a reduced level of severe toxicity compared to those at the median dose. These findings have led to the design of a study with the goal of reducing high levels of toxicity in sarcopenic patients. If the expected level of dose limiting toxicity in sarcopenic patients is 80% based on the standard method of dosing, this could be expected to be reduced to the median value of 41% dose limiting toxicity by the administration of cisplatin scaled to individual lean body mass. Hypothesis: Levels of severe toxicity in sarcopenic patients may be reduced to clinically acceptable levels by cisplatin dosing scaled to 3.1 mg/kg lean body mass compared with standard dosing of 75 mg/m2 based on body surface area.

ELIGIBILITY:
Inclusion Criteria:

* Recommendation from treating oncologist to receive a cisplatin based chemotherapy regimen, specifically either cisplatin/vinorelbine or cisplatin/gemcitabine
* > or = 18 years of age
* Histologically proven diagnosis of non-small cell lung cancer, Stage IIIB or IV
* Adequate renal function: creatinine < 1.5 mg/dL or < 132 µmol/L and creatinine clearance of > 45 mL/min using the Cockcroft-Gault formula
* Adequate hepatic function: bilirubin < 1.5 mg/dL or < 25 µmol/L and AST and ALT < 2 times upper limit of normal, unless there is evidence of liver metastases, in which case < 5 times upper limit of normal
* Adequate hematological function: absolute neutrophil count (ANC) > 1.5 x 109/L and platelets > 100 x 109/L and hemoglobin > 100 g/L
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Negative serum pregnancy test for women of childbearing potential. Women and men of child bearing potential must use effective contraception defined as the simultaneous use of two reliable methods unless abstinence is the chosen method.
* Life expectancy of > 4 months in the opinion of the treating oncologist
* Prior radiotherapy is allowed (unless > 25% of bone marrow stores) if this radiation was > 4 weeks before study entry and patient has fully recovered from toxicity of this treatment
* Willingness to comply with the study protocol
* Ability to give written informed consent with the understanding that it may be withdrawn at any time without prejudice

Exclusion Criteria:

* Pregnant or lactating women
* Brain metastases (a CT or MRI is not required to rule out brain metastases unless there is clinical suspicion)
* Previous or concurrent malignancies, excluding curatively treated in situ carcinoma of the cervix, in situ ductal breast cancer, non-melanoma skin cancer or low grade bladder cancer
* Patients who have had major surgery within three weeks of enrollment without a full recovery
* Prior treatment with any anticancer therapy
* Patients who have tested positive for HIV
* Any significant medical or psychiatric condition that, in the opinion of the investigator, will exclude the patient from the study for compliance or safety reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity rates | Assessed weekly until patients come off study (an expected average of 9 weeks)
Number of Cycles completed | Assessed weekly until patients come off study (an expected average of 9 weeks)

SECONDARY OUTCOMES:
Survival | Assessed every 60 days from the date of removal from the trial (an expected average of 9 months)
  If a patient has deceased, the date of death is recorded. If a patient is alive, the status is checked again in another 60 days. This is carried out through health records and not through direct contact with the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Sawyer, MD, Principal Investigator — Medical Oncologist, Cross Cancer Institute; Vickie Baracos, PhD, Study Chair — Grant Holder, Department of Oncology, University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Prado CM, Lieffers JR, McCargar LJ, Reiman T, Sawyer MB, Martin L, Baracos VE. Prevalence and clinical implications of sarcopenic obesity in patients with solid tumours of the respiratory and gastrointestinal tracts: a population-based study. Lancet Oncol. 2008 Jul;9(7):629-35. doi: 10.1016/S1470-2045(08)70153-0. Epub 2008 Jun 6. PMID 18539529
- [Background] Tan BH, Birdsell LA, Martin L, Baracos VE, Fearon KC. Sarcopenia in an overweight or obese patient is an adverse prognostic factor in pancreatic cancer. Clin Cancer Res. 2009 Nov 15;15(22):6973-9. doi: 10.1158/1078-0432.CCR-09-1525. Epub 2009 Nov 3. PMID 19887488
- [Background] Prado CM, Baracos VE, McCargar LJ, Mourtzakis M, Mulder KE, Reiman T, Butts CA, Scarfe AG, Sawyer MB. Body composition as an independent determinant of 5-fluorouracil-based chemotherapy toxicity. Clin Cancer Res. 2007 Jun 1;13(11):3264-8. doi: 10.1158/1078-0432.CCR-06-3067. PMID 17545532
- [Background] Prado CM, Baracos VE, McCargar LJ, Reiman T, Mourtzakis M, Tonkin K, Mackey JR, Koski S, Pituskin E, Sawyer MB. Sarcopenia as a determinant of chemotherapy toxicity and time to tumor progression in metastatic breast cancer patients receiving capecitabine treatment. Clin Cancer Res. 2009 Apr 15;15(8):2920-6. doi: 10.1158/1078-0432.CCR-08-2242. Epub 2009 Apr 7. PMID 19351764
- [Background] Antoun S, Birdsell L, Sawyer MB, Venner P, Escudier B, Baracos VE. Association of skeletal muscle wasting with treatment with sorafenib in patients with advanced renal cell carcinoma: results from a placebo-controlled study. J Clin Oncol. 2010 Feb 20;28(6):1054-60. doi: 10.1200/JCO.2009.24.9730. Epub 2010 Jan 19. PMID 20085939